CLINICAL TRIAL: NCT01885741
Title: A Prospective, Open-Label, Single-Arm, Single-Site, Study to Demonstrate the Preliminary Safety and Effectiveness of IPBS in Performing MRI-Guided Targeting and Intervention of Breast Tissue in Female Patients Indicated for MRI-Guided Breast Biopsy.
Brief Title: Study to Demonstrate the Preliminary Safety and Effectiveness of IPBS in Performing MRI-Guided Targeting and Intervention of Breast Tissue in Female Patients Indicated for MRI-Guided Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IPBS-001
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer Screening; MRI Guided Breast Biopsy; Breast Cancer Diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPBS (Experimental)
  Interventions: Device: IPBS

INTERVENTIONS:
Device: IPBS

SUMMARY:
A preliminary demonstration of the Safety of IPBS in positioning a vacuum assisted biopsy (VAB) tool to enable an MRI-guided automated breast biopsy. This will consist of 10-15 biopsy procedures facilitated by the MRI-guided system. Patients will be followed after the procedure to assess clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 18 with suspected or confirmed breast cancer requiring a manual MRI-guided breast biopsy for diagnosis and staging.
* Individuals Capable of giving a free and informed consent.

Exclusion Criteria:

* Any patient for whom the manual MRI-guided breast biopsy procedure would not be possible (size of patient, etc.).
* Patients who refuse the procedure for any reason will be excluded from the study at the investigators discretion.
* Patients who are not suitable for the procedure will be excluded at the investigators discretion.
* Patients unwilling to complete associated study questionnaires or follow up visits.
* Women who are pregnant or who plan to become pregnant within the study duration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Frequency of target reached by the interventional tools as determined by a qualified physician reviewing the MR images. | Day 1

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hopital du Saint-Sacrement, Québec, Quebec